CLINICAL TRIAL: NCT05497531
Title: Pilot Trial Comparing Circulating Tumor DNA (ctDNA) From Immediate Draining Vein vs. Standard Peripheral Vein Sample in Patients Undergoing Biopsies for Hepatobiliary and Pancreatic Cancers
Brief Title: Pilot Comparing ctDNA IDV vs. SPV Sample in Pts Undergoing Biopsies for Hepatobiliary and Pancreatic Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Nadine Abi-Jaoudeh, Professor of Radiological Sciences, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1491; UCI 21-124 (Other: UCI CFCCC)
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Hepatobiliary Cancer; Pancreatic Cancer; Hepatocellular Carcinoma; Cholangiocarcinoma; Ampullary Cancer; Pancreatic Carcinoma
Keywords: ctDNA; Circulating Tumor DNA; Pancreatic Cancer; Hepatobiliary Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ctDNA collection from draining and peripheral veins (Experimental): Patient with suspected primary hepatobiliary or pancreatic cancer undergoing a diagnostic work-up with a percutaneous or trans-jugular biopsy (standard of care) and will undergo a sampling of the cancer draining vein during their biopsy procedure with a collection of an additional 10mL of blood.
  Interventions: Diagnostic Test: ctDNA Blood Collection

INTERVENTIONS:
Diagnostic Test: ctDNA Blood Collection — Blood collection to be obtained from peripheral vein and cancer draining vein during biopsy

SUMMARY:
This is a prospective pilot protocol investigating whether ctDNA detection be improved by sampling the cancer draining vein versus the standard practice of sampling from a peripheral vein in patients who are undergoing biopsies for hepatobiliary and pancreatic cancers.

DETAILED DESCRIPTION:
This is a, prospective single center pilot study to investigate whether ctDNA detection can be improved by sampling the cancer draining vein vs. a peripheral vein (current practice). As a secondary endpoint, both ctDNA results will be compared with percutaneous biopsy (standard of care).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have or are undergoing work-up for hepatobiliary and/or pancreatic carcinoma (such as hepatocellular carcinoma, cholangiocarcinoma, ampullary carcinoma, pancreatic carcinoma)
* Scheduled for an image-guided percutaneous or trans-jugular biopsy of a lesion
* Must be able to provide a written informed consent

Exclusion Criteria:

* Patients unable to hold reasonably still on a procedure table or hold their breath during imaging or needle passes
* Patients with a gross body weight over 375 pounds (upper limit of the CT and angiography tables)
* Patients with uncorrectable coagulopathy
* Platelet count < 30,000/ul
* International Normalized (INR) > 1.5
* Patients with moderate to severe ascites who cannot undergo trans-jugular biopsy or sufficient drainage
* No clear reachable target for percutaneous or trans-jugular biopsy
* Patient who cannot have a peripheral blood draw for ctDNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the amount of ctDNA in draining vein plasma sample to peripheral vein sample through ratio of mean allele frequency | Up to 1 year
  Ratio of mean allele frequency (MAF)% of hepatic or portal draining vein, and MAF% of peripheral blood will be utilized to compare the samples

SECONDARY OUTCOMES:
Number of unique alterations found in hepatic or portal vein plasma compared to number of alterations found in peripheral vein plasma | Up to 1 year
  ctDNA results will be compared with percutaneous biopsy (standard of care)
Number of unique alterations found in ctDNA compared to number of alterations derived next generation sequencing (NGS) | Up to 1 year
  ctDNA results will be compared with percutaneous biopsy (standard of care)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Abi-Jaoudeh, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States